CLINICAL TRIAL: NCT03520231
Title: A Multicenter Randomized Double Blind Study Examining the Efficacy and Safety of Denosumab in Combination With First Line Platinum-based Chemotherapy for Patients With Bone Metastasis Secondary to Metastatic Urothelial Cancer
Brief Title: Study Comparing Denosumab With Standard Treatment in Urothelial Cancer Patients With Bone Metastases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DENIM
Record Dates: First submitted 2018-04-27; First posted 2018-05-09 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2020-09

CONDITIONS: Urothelial Carcinoma; Kidney Cancer; Ureter Cancer; Bladder Cancer
MeSH Terms: conditions — Carcinoma, Transitional Cell; Kidney Neoplasms; Ureteral Neoplasms; Urinary Bladder Neoplasms | interventions — Denosumab; Gemcitabine; Carboplatin; Cisplatin; Calcium; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Denosumab and Standard Chemotherapy (Experimental): Denosumab, given subcutaneously at a dose of 120 mg, every 4 weeks.
  Gemcitabine, given intravenously at standard doses, on Days 1 and 8 of every 21 day cycle, for 3-4 cycles.
  Carboplatin, given intravenously at standard doses, on Day 1 of every 21 day cycle, for 3-4 cycles.
  OR Cisplatin, given intravenously at standard doses, on Day 1 of every 21 day cycle, for 3-4 cycles.
  Calcium, orally at a dose of 1000 mg, once daily.
  Vitamin D, orally at a dose of 400 IU, once daily.
  Interventions: Drug: Denosumab; Drug: Gemcitabine; Drug: Carboplatin; Drug: Cisplatin; Dietary Supplement: Calcium; Dietary Supplement: Vitamin D
- Denosumab Placebo and Standard Chemotherapy (Placebo Comparator): Denosumab placebo, given subcutaneously, every 4 weeks.
  Gemcitabine, given intravenously at standard doses, on Days 1 and 8 of every 21 day cycle, for 3-4 cycles.
  Carboplatin, given intravenously at standard doses, on Day 1 of every 21 day cycle, for 3-4 cycles.
  OR Cisplatin, given intravenously at standard doses, on Day 1 of every 21 day cycle, for 3-4 cycles.
  Calcium, orally at a dose of 1000 mg, once daily.
  Vitamin D, orally at a dose of 400 IU, once daily.
  Interventions: Other: Denosumab Placebo; Drug: Gemcitabine; Drug: Carboplatin; Drug: Cisplatin; Dietary Supplement: Calcium; Dietary Supplement: Vitamin D

INTERVENTIONS:
Drug: Denosumab — RANK Ligand Inhibitor
  Other Names: XGEVA
  Arms: Denosumab and Standard Chemotherapy
Other: Denosumab Placebo — Placebo
  Arms: Denosumab Placebo and Standard Chemotherapy
Drug: Gemcitabine — Antineoplastic Agent
Drug: Carboplatin — Antineoplastic Agent
Drug: Cisplatin — Antineoplastic Agent
Dietary Supplement: Calcium — Calcium Supplement
Dietary Supplement: Vitamin D — Vitamin D Supplement

SUMMARY:
This is a phase 2 study of the drug denosumab for the management bone metastases from urothelial cancer.

The purpose of this study is to find out how effective denosumab is in the management of bone metastases from urothelial cancer. This will be done by comparing denosumab with standard treatment, compared to placebo and standard treatment.

Denosumab is a monoclonal antibody that binds to a protein called Receptor Activator of Nuclear Factor κB (RANK). RANK works by telling certain cells called osteoclasts to break down bone tissue. The binding of denosumab to RANK stops it from telling osteoclasts to break down bone tissue which may help with symptoms related bone metastases from urothelial cancer.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double blind, Phase II study. Participants eligible for this study have metastatic urothelial cancer and bone metastases and are planned to receive 4-6 cycles of a standard of care platinum-doublet regimen. In a double blind manner, 50 participants will be randomized in a 1:1 ratio to receive denosumab 120 mg or matching placebo subcutaneously every 4 weeks with their first dose coinciding with the first cycle of chemotherapy. Patients will continue on denosumab/placebo even after all planned chemotherapy cycles have been delivered and until the end of the study at 18 months after the last dose of chemotherapy. Patients with symptomatic progression in the bone may be unblinded and crossed over to denosumab (if on placebo). All participants will be provided with 1000 mg of calcium and 400 IU of vitamin D to be taken daily. Participants who discontinue the investigational product early will be followed for disease status and survival.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed urothelial carcinoma (kidney, ureter, bladder) with metastatic disease involving the bones, not amenable to curative treatment
* Mixed histologies permitted as long as urothelial histology is the major component Presence of one or more bone metastases
* No prior systemic chemotherapy for metastatic disease (immunotherapy permitted)
* Starting first line chemotherapy for metastatic urothelial cancer with gemcitabine and cisplatin or gemcitabine and carboplatin and planned to receive 4-6 cycles
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Adequate renal function
* Acceptable serum calcium or albumin-adjusted serum calcium
* Adequate hepatic function
* Patients all require oral examination and appropriate preventative dentistry prior to starting treatment
* Expected life expectancy of at least 3 months

Exclusion Criteria:

* Prior chemotherapy for metastatic disease
* Current or prior IV bisphosphonate or denosumab administration
* Current or prior oral bisphosphonate administration to treat bone metastases
* Unacceptable renal function
* Abnormal bone metabolism (Paget's disease)
* Untreated or symptomatic brain metastases
* Patients with a history of other malignancies, with exceptions
* Significant dental/oral disease
* Administration of other prior anticancer therapies within 2 weeks of randomization
* Patient is pregnant or breast feeding, or planning to become pregnant within 7 months after the end of treatment
* Female of child bearing potential is not willing to use, in combination with her partner, highly effective contraception during treatment and for 7 months after the end of treatment
* Known sensitivity to any of the products to be administered during the study
* History of any other clinically significant disorder, condition or disease that in the opinion of the investigator excludes the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Difference in mean percentage change in serum c-telopeptide (sCTX) between the two arms (investigational drug arm and placebo arm). | Baseline to Week 10
  Mean percentage change should be greater than or equal to 30%.

SECONDARY OUTCOMES:
Number of patients with a change in sCTx | Baseline to Week 10
  To determine the proportion of patients with a change in sCTx of >30% from baseline at week 1 to week 10
Mean percentage change in serum bone-specific alkaline phosphatase (bALP) in the investigational arm | Baseline to Week 10
Mean percentage change in urinary N-telopeptide (uNTx) levels in the investigational arm | Baseline to Week 10
Mean percentage change in sCTx levels in the investigational arm | Baseline to End of Chemotherapy (Week 20)
Mean percentage change in bALP levels in the investigational arm | Baseline to End of Chemotherapy (Week 20)
Mean percentage change in uNTx levels in the investigational arm | Baseline to End of Chemotherapy (Week 20)
Mean percentage change in serum bone-specific alkaline phosphatase (bALP) in the placebo arm. | Baseline to Week 10
Mean percentage change in urinary N-telopeptide (uNTx) levels in the placebo arm. | Baseline to Week 10
Mean percentage change in sCTx levels in the levels in the placebo arm. | Baseline to End of Chemotherapy (Week 20)
Mean percentage change in bALP levels in the levels in the placebo arm. | Baseline to End of Chemotherapy (Week 20)
Mean percentage change in uNTx levels in the levels in the placebo arm. | Baseline to End of Chemotherapy (Week 20)
Time to first on study symptomatic skeletal related events | 2 years
  To determine and compare the time to first on study symptomatic skeletal related events (SSE); (fracture, surgery, radiation to bone, or spinal cord compression) between each arm of the study
Progression free survival rate | 1 year
  To determine progression free survival (PFS) in each arm at 1 year (with appropriate censoring) after last dose of chemotherapy
Progression free survival rate | 18 months
  To determine progression free survival (PFS) in each arm at 18 months (with appropriate censoring) after last dose of chemotherapy
Overall survival rate | 1 year
  To determine overall survival (OS) rate at 1 year (with appropriate censoring) after last dose of chemotherapy
Overall survival rate | 18 months
  To determine overall survival (OS) rate at 18 months (with appropriate censoring) after last dose of chemotherapy
Number of participants with side effects in the investigational drug arm | 2 years
  To evaluate safety and tolerability
Number of participants with side effects in the placebo arm | 2 years
  To evaluate safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Srikala Sridhar, M.D., Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No